CLINICAL TRIAL: NCT06830083
Title: Hypofractionated Radiation Fractionation in Breast Cancer Patients with Implant-Based Reconstruction
Acronym: HFIBR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Jiangsu Taizhou People's Hospital (Other); Hunan Cancer Hospital (Other)
Responsible Party: Principal Investigator, Sun Xinchen, The First Affiliated Hospital of Nanjing Medical University (Jiangsu Provincial People's Hospital), The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: First Affiliated Hospital, Nan
Record Dates: First submitted 2025-01-26; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: implant-based reconstruction surgery; hypofraction radiation therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- conventional fraction radiotherapy (Active Comparator): Total dose of plan tumor volume is 5000 cGy，and each fraction will consist of 200 cGy per day. 25 fractions(daily, Monday through Friday) to the chest wall and to the regional (with or without axillary) lymph nodes.
  Interventions: Radiation: Conventional fraction radiotherapy
- hypofractioned radiotherapy (Experimental): Total dose of plan tumor volume is 4050 cGy，and each fraction will consist of 270 cGy per day. 15 fractions(daily, Monday through Friday) to the chest wall and to the regional (with or without axillary) lymph nodes.
  Interventions: Radiation: Hypofractionated Radiation Therapy

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Hypofractionation regimen: Total dose to the chest wall and the regional lymph nodes is 4050 cGy, and each fraction consists of 270 cGy per day(daily, Monday through Friday )
  Other Names: HF
  Arms: hypofractioned radiotherapy
Radiation: Conventional fraction radiotherapy — Total dose of plan tumor volume is 5000 cGy，and each fraction will consist of 200 cGy per day. 25 fractions(daily, Monday through Friday) to the chest wall and to the supraclavicular (with or without axillary) lymph nodes.
  Other Names: CF
  Arms: conventional fraction radiotherapy

SUMMARY:
It is a randomized trial to assess the safety and efficacy between hypofractionation radiation and conventional radiation in women who have undergone mastectomy and immediate breast reconstruction. The investigators will evaluate reconstruction complication, radiotherapy side effects, cosmetic and oncologic outcomes.

DETAILED DESCRIPTION:
Patients with breast cancer frequently have requirement for breast reconstruction after mastectomy. For patients with limited autologous tissue availability, implant-based reconstruction remains an effective alternative. Due to the absence of high-level evidence, collaborative efforts between surgical and radiation oncology teams are advised to determine the optimal sequencing and techniques for integrating reconstruction surgery with radiotherapy. The ongoing Alliance A221505 and FABREC phase III randomized controlled trials are comparing the incidence of reconstructive complications following hypofractionated and conventional fractionation radiotherapy. FABREC trial recently showed the hypofractionated regimen did not significantly improve change in physical well-being（PWB), domain of the Functional Assessment of Cancer Therapy-Breast (FACT-B) quality-of-life assessment tool, compared with the conventional fractionation radiotherapy. This trial added to the increasing experience with HF PMRT in patients with implant-based reconstruction.

In 2019, the European Society for Radiotherapy and Oncology (ESTRO) provided guidelines for target delineation based on the position of the implant in breast reconstruction to minimize the irradiation of normal tissues. Existing studies on the risk of complications from irradiating expanders and implants have yielded inconsistent conclusions, with each approach having its own advantages and disadvantages.

Our study aims to compare the incidence of reconstructive complications between hypofractionated and conventional fractionation radiotherapy after implant-based reconstruction surgery to provide high-level evidence for medium-dose hypofractionated radiotherapy after immediate implant-based reconstructive surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis of stage I-III breast cancer (non-T4), >18 years old; 2. Complete breast cancer resection (including skin-sparing and nipple-sparing total resection) 3. According to the guidelines of the Chinese Anticancer Society, postoperative adjuvant radiotherapy is required; 4. Undergo immediate reconstructive surgery (tissue dilator or permanent implant)

Exclusion Criteria:

1. Auto-reconstruction surgery
2. Clinical or pathological T4
3. Both sides need radiotherapy
4. Have a history of chest radiotherapy
5. Pregnancy/lactation
6. Participate in other drug clinical trials

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 840 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Major complication | From enrollment to the end of treatment at 24 months
  implant related complications requiring reoperation such as severe necrosis，severe infections, severe capsular contracture, implant rupture and implant exposure.

SECONDARY OUTCOMES:
Any breast-related complications | From enrollment to the end of treatment at 24 months
  Complications included infections, wound dehiscence, skin flap necrosis, implant exposure, capsular contracture, seroma, and hematoma.
Absolute reconstruction failure | From enrollment to the end of treatment at 24 months
Oncologic outcomes | From enrollment to the end of treatment at 5 years
  local-regional recurrence free survival
Cosmetic outcomes | From enrollment to the end of treatment at 24 months
  satisfaction with breast and physical and psychosocial well-bing after radiotherapy will be assessed from baseline to 24 months by trained physicians using Breast-Q Version 2.0© Reconstruction Module Scales Chinese (CN) Version .

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province People's Hospital/The First Affiliated with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mutter RW, Giri S, Fruth BF, Remmes NB, Boughey JC, Harless CA, Ruddy KJ, McGee LA, Afzal A, Gao RW, Shumway DA, Vern-Gross TZ, Villarraga HR, Kenison SL, Kang Y, Wong WW, Stish BJ, Merrell KW, Yan ES, Park SS, Corbin KS, Vargas CE. Conventional versus hypofractionated postmastectomy proton radiotherapy in the USA (MC1631): a randomised phase 2 trial. Lancet Oncol. 2023 Oct;24(10):1083-1093. doi: 10.1016/S1470-2045(23)00388-1. Epub 2023 Sep 8. PMID 37696281
- [Background] Wong JS, Uno H, Tramontano AC, Fisher L, Pellegrini CV, Abel GA, Burstein HJ, Chun YS, King TA, Schrag D, Winer E, Bellon JR, Cheney MD, Hardenbergh P, Ho A, Horst KC, Kim JN, Leonard KL, Moran MS, Park CC, Recht A, Soto DE, Shiloh RY, Stinson SF, Snyder KM, Taghian AG, Warren LE, Wright JL, Punglia RS. Hypofractionated vs Conventionally Fractionated Postmastectomy Radiation After Implant-Based Reconstruction: A Randomized Clinical Trial. JAMA Oncol. 2024 Oct 1;10(10):1370-1378. doi: 10.1001/jamaoncol.2024.2652. PMID 39115975
- [Background] Wang SL, Fang H, Song YW, Wang WH, Hu C, Liu YP, Jin J, Liu XF, Yu ZH, Ren H, Li N, Lu NN, Tang Y, Tang Y, Qi SN, Sun GY, Peng R, Li S, Chen B, Yang Y, Li YX. Hypofractionated versus conventional fractionated postmastectomy radiotherapy for patients with high-risk breast cancer: a randomised, non-inferiority, open-label, phase 3 trial. Lancet Oncol. 2019 Mar;20(3):352-360. doi: 10.1016/S1470-2045(18)30813-1. Epub 2019 Jan 30. PMID 30711522
- [Background] Salvestrini V, Valzano M, Meattini I, Becherini C, Visani L, Francolini G, Morelli I, Bertini N, Orzalesi L, Bernini M, Bianchi S, Simontacchi G, Livi L, Desideri I. Anatomical assessment of local recurrence site in breast cancer patients after breast reconstruction and post-mastectomy radiotherapy: implications for radiation volumes and techniques. Radiol Med. 2024 Jun;129(6):845-854. doi: 10.1007/s11547-024-01812-z. Epub 2024 Apr 11. PMID 38602657
- [Background] Wu ZY, Han HH, Kim HJ, Lee J, Chung IY, Kim J, Lee S, Han J, Eom JS, Kim SB, Gong G, Kim HH, Son BH, Ahn SH, Ko B. Locoregional recurrence following nipple-sparing mastectomy with immediate breast reconstruction: Patterns and prognostic significance. Eur J Surg Oncol. 2021 Jun;47(6):1309-1315. doi: 10.1016/j.ejso.2021.01.006. Epub 2021 Jan 13. PMID 33495030
- [Background] Kaidar-Person O, Vrou Offersen B, Hol S, Arenas M, Aristei C, Bourgier C, Cardoso MJ, Chua B, Coles CE, Engberg Damsgaard T, Gabrys D, Jagsi R, Jimenez R, Kirby AM, Kirkove C, Kirova Y, Kouloulias V, Marinko T, Meattini I, Mjaaland I, Nader Marta G, Witt Nystrom P, Senkus E, Skytta T, Tvedskov TF, Verhoeven K, Poortmans P. ESTRO ACROP consensus guideline for target volume delineation in the setting of postmastectomy radiation therapy after implant-based immediate reconstruction for early stage breast cancer. Radiother Oncol. 2019 Aug;137:159-166. doi: 10.1016/j.radonc.2019.04.010. Epub 2019 May 17. PMID 31108277
- [Background] Kim YH, Yang YJ, Lee DW, Song SY, Lew DH, Yang EJ. Prevention of Postoperative Complications by Prepectoral versus Subpectoral Breast Reconstruction: A Systematic Review and Meta-Analysis. Plast Reconstr Surg. 2024 Jan 1;153(1):10e-24e. doi: 10.1097/PRS.0000000000010493. Epub 2023 Apr 4. PMID 37010460
- [Background] Zhang X, Ning S, Zhang Y. Complications After Prepectoral Versus Subpectoral Breast Reconstruction in Patients Receiving Postmastectomy Radiation Therapy: A Systematic Review and Meta-Analysis. Aesthetic Plast Surg. 2024 Nov;48(21):4421-4429. doi: 10.1007/s00266-024-04096-w. Epub 2024 May 3. PMID 38700543
- [Background] Jagsi R, Momoh AO, Qi J, Hamill JB, Billig J, Kim HM, Pusic AL, Wilkins EG. Impact of Radiotherapy on Complications and Patient-Reported Outcomes After Breast Reconstruction. J Natl Cancer Inst. 2018 Feb 1;110(2):157-65. doi: 10.1093/jnci/djx148. PMID 28954300